CLINICAL TRIAL: NCT00500201
Title: A Single Blind, Double Dummy, Placebo Controlled, Randomized, 2 Period Crossover Study to Assess the Relative Bioavailability of a 120mg Tablet Compared to Two 60 mg SB-773812 Tablets in Healthy Volunteers
Brief Title: A Healthy Volunteer Study to Assess the Relative Bioavailability of 2 Forms of SB773812 Tablets.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: NAA105737
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
Keywords: Healthy Volunteer
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects in treatment sequence AB (Experimental): In treatment sequence AB first subjects will be randomized to receive treatment A (two tablets of 60 milligram [mg] of SB-773812) and one placebo tablet. Then subjects will receive treatment B (one tablet of 120 mg of SB-773812) and two placebo tablets . There will be a wash-out period of 20 days between.
  Interventions: Drug: SB- 773812 60 mg; Drug: SB- 773812 120 mg; Drug: Placebo
- Subjects in treatment sequence BA (Experimental): In treatment sequence BA first subjects will be randomized to receive treatment B (one tablet of 120 mg of SB-773812) and two placebo tablets. Then subjects will receive treatment A (two tablets of 60 mg of SB-773812) and one placebo tablet. There will be a wash-out period of 20 days between.
  Interventions: Drug: SB- 773812 60 mg; Drug: SB- 773812 120 mg; Drug: Placebo

INTERVENTIONS:
Drug: SB- 773812 60 mg — SB- 773812 will be available dose strength of 60 mg and administered orally by subjects.
  Other Names: SB- 773812
Drug: SB- 773812 120 mg — SB- 773812 will be available dose strength of 120 mg and administered orally by subjects.
Drug: Placebo — Placebo tablets will be administered orally by subjects.

SUMMARY:
Study to compare PK of a new 120mg tablet with two 60mg tablets. This is required because we plan to have only single tablets administered in the later phase clinical trials but we have not had a 120mg strength before. As this is a new previously untested strength we need to ensure that the PK is similar to that achieved using 2x60mg before we start a large manufacturing campaign and before we administer to a large number of patients. The study is planned to consist of a single part, with two dosing periods, periods 1 and 2 consisting of 18 subjects. There will be 20 days washout between each dose. Initially 4 subjects will be given a single oral dose of 120 mg SB-773812 and 2 will be given placebo. If 120mg SB-773812 is well tolerated in the first four volunteers, the remaining 12 subjects will be dosed. If the 120mg single oral dose in the first 4 subjects is poorly tolerated, the study will be stopped. Subjects will return to the centre for follow-up 14 to 21 days after the final dose.It is expected that the total duration of the study should be approximately 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* be a healthy man or woman, aged 18 to 55, and be neither too fat nor too thin;
* If you are a woman who can have a baby, you must use an acceptable method of contraception, from the start of your last period before you take the study medicine, until you've had your first normal period after the end of the study. You might need to use contraception for longer than that. You don't need to use contraception if your partner has been sterilized (had an operation to cut the tubes that carry sperm).
* Acceptable methods of contraception for women are:
* Diaphragm or cap and condom with spermicide;
* the 'Pill' and condom with spermicide - you must have been taking the 'Pill' for at least 3 months before the start of the study;
* Intrauterine device (IUD or 'coil' - your GP must confirm that you have one) and condom with spermicide; or
* Condom and spermicide only, if you're a woman who has had an operation to have your tubes tied.
* If you are a woman who CANNOT have a baby, you should have gone through menopause at least 1 year ago;
* had your womb removed; or
* had both ovaries removed.
* have normal physical exam
* have normal blood pressure and pulse.
* be able to swallow tablets;
* show proof of identity - we'll tell you what's suitable.
* have the ability to understand and comply with protocol requirements, instructions and restrictions.
* be available to attend the ward for repeat tests, if necessary, during the 2 weeks after your final planned visit.

Exclusion Criteria:

* abuse alcohol or drugs;
* drink, on average, more than 3 units of alcohol daily if you're a man, or 2 units if you're a woman (1 unit = ½ pint of beer, 1 small glass of wine or 1 measure of spirits);
* have been a blood donor in the last 3 months;
* have been given an experimental medicine in the last 3 months;
* have taken part in a study of an experimental medicine in the last 3 months;
* be a smoker, or have smoked cigarettes or used other tobacco products regularly in the last 6 months - we may test your breath for smoking at any time during the study;
* be pregnant or breast feeding;
* have had a serious reaction to any medicine;
* have any screening test results that show you're not suitable, even if they don't mean that you're unhealthy;
* have had any important illness (including diabetes and asthma) that, in the opinion of the study doctor, makes you unsuitable for the study;
* have had any mental illnesses;
* suffer from numbness or tingling in your arms, legs, hands or feet; or
* has had glaucoma (increased pressure inside the eye).
* You may not be able to take part if you've taken any medicines recently, including herbal remedies like St John's wort.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05-24 (Actual); Primary Completion 2007-07-25 (Actual); Study Completion 2007-07-25 (Actual)

PRIMARY OUTCOMES:
Blood sampling over a period 336 hrs post SB773812 dosing in both dosing sessions. | 336 hrs post SB773812 dosing

SECONDARY OUTCOMES:
Safety: ECG, vital signs, clinical labs over 336 hours post SB-773812 dosing in both dosing sessions. | 336 hours post SB-773812 dosing
Continuous adverse event monitoring from dosing until study conclusion and follow up, 7-14days after last dose. | 7-14days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study NAA105737 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/NAA105737?search=study&search_terms=NAA105737#rs